CLINICAL TRIAL: NCT04973618
Title: Phase 1B Study of APVO436 in Combination With Venetoclax and Azacitidine in Elderly or Unfit Patients With Newly Diagnosed Acute Myeloid Leukemia (AML)
Brief Title: Study of APVO436 in Elderly or Unfit Patients With Newly Diagnosed AML
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Change of strategy
Sponsor: Aptevo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5002
Record Dates: First submitted 2021-07-12; First posted 2021-07-22 (Actual); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: AML
Keywords: APVO436

STUDY DESIGN:
Intervention Model Description: APVO436 will be administered at a fixed dosage of 18 mcg after a weekly ramp up during Cycle 1 (Step-up dosing: C1D15: 6 mcg over 22 hours, C1D22: 12 mcg over 8 hours, C2D1: 18 mcg over 6 hours, C2D8: 18 mcg over 4 hours), totaling 18 µg in Cycle 1 and 72 µg/cycle for Cycles 2-4 for a total of 234 µg for the projected 4-cycle treatment course.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- APVO436 (Experimental): CD123 and CD3 epsilon bispecific antibody
  Interventions: Biological: APVO436

INTERVENTIONS:
Biological: APVO436 — APVO436
  Dosage: APVO436 will be administered at a fixed dosage of 18 mcg after a weekly ramp up during Cycle 1 (Step-up dosing: C1D15: 6 mcg over 22 hours, C1D22: 12 mcg over 8 hours, C2D1: 18 mcg over 6 hours, C2D8: 18 mcg over 4 hours), totaling 18 µg in Cycle 1 and 72 µg/cycle for Cycles 2-4 for a total of 234 µg for the projected 4-cycle treatment course.
  Dosage Form: IV Solutions for Intravenous Administration
  Frequency: Weekly

SUMMARY:
The goal of this Phase IB study is to evaluate the safety and tolerability of APVO436 in naïve elderly unfit patients with newly diagnosed primary AML at the RP2D level when it is used as an adjunct to the standard of care and obtain a preliminary assessment of the anti-leukemia activity of an APVO436-containing combination therapy.

Study Objectives:

- Primary Objective: Evaluate the safety and tolerability of APVO436 at the RP2D level when it is used as an adjunct to the standard of care (venetoclax and azacitidine).

- Secondary Objectives:

* Obtain a preliminary assessment of the anti-leukemia activity of APVO436-containing experimental triple drug combination therapy modalities.
* Determine pharmacodynamics (PD) of APVO436, including changes in CD123 antigen density and measures of T cell number and function over time.
* Determine correlations between response and MRD level and cytogenetic and molecular genetic profiles.

DETAILED DESCRIPTION:
The goal of this Phase IB study is to evaluate the safety and tolerability of APVO436 at the RP2D level when it is used as an adjunct to the standard of care and obtain a preliminary assessment of the anti-leukemia activity of an APVO436-containing combination therapy.

The MTD for APVO436 was not reached at a dose level of 240 µg/cycle in the ongoing Phase 1 FIHT (Cohort 10 in the dose escalation phase; weekly dose 60 mcg). 46 patients have received intravenous infusions of APVO436 across multiple dose-escalation cohorts, with dosing escalated from 0.3 micrograms to 60 micrograms. Long half-life of APVO436 enabled its administration over short infusion times. APVO436 exhibited a manageable safety profile, encouraging single agent activity and a promising benefit to risk profile in relapsed advanced stage AML. Of 7 evaluable relapsed AML patients treated in Cohort 6, 5 showed stabilization of their leukemia. Of the 5 AML patients with disease stabilization, 3 lived 246+ days, 261+ days, and 281+ days, respectively and 2 progressed after a month. Two of the patients who experienced a stabilization of their relapsed leukemia achieved first a partial remission (PR) and subsequently a complete remission (CR). No partial or complete remissions were observed at APVO436 dose levels lower or higher than the Cohort 6 dose level. The sub-MTD dose level of Cohort 6 was identified as the RP2D level of APVO436 for further evaluation in this study. Therefore, APVO436 will be used at the Cohort 6 dose level from Study 5001 in this study. CRS has occurred in some patients and has been managed using the generally recommended standard CRS treatments". In Cohort 6, among 9 AML/MDS patients evaluable for toxicity, 2 patients developed a Grade 1 CRS and one patient developed a transient Grade 3 CRS related to APVO436 which resolved with routine clinical management.

A total of 20 eligible patients will be enrolled in the current study. APVO436 will be administered intravenously over 4 hours weekly on days 1, 8, 15, and 22 of each cycle at a fixed dosage of 18 mcg after a weekly ramp up during Cycle 1 (Step-up dosing: C1D15: 6 mcg over 22 hours, C1D22: 12 mcg over 8 hours, C2D1: 18 mcg over 6 hours, C2D8: 18 mcg over 4 hours). The infusion time may be increased to 22 hours if deemed appropriate and/or necessary by the PI.

Patients will receive 4 x 28-day cycles of combined 3-drug immunochemotherapy: APVA [APVO436+Venetoclax+Azacitidine]

Optional continued triple therapy for 4 additional cycles (up to 8 total cycles) will be available for patients with an objective working group response or prolonged stable disease/clinical benefit. Patients completing 8 cycles of triple therapy on protocol will then move to follow-up and continue SOC therapy per their treating physician.

Venetoclax will be administered orally daily on days 1-21 of each cycle at a fixed dosage of 400 mg/daily after a daily ramp up (Day 1: 100 mg; Day 2: 200 mg; Day 3-Day 21: 400 mg). Standard dose adjustments will be made for patients on azole antifungals.

Azacitidine will be administered intravenously over 30 min daily on days 1-7 of each cycle at a dosage of 75 mg/m2

ELIGIBILITY:
Inclusion Criteria:

Individuals eligible to participate in this study must meet all of the following:

All patients must meet the following criteria prior to the first dose of study drug:

1. Signed informed consent. Consent must be obtained prior to any study-related procedure.
2. Age ≥60 years
3. Histologically confirmed AML: Subjects must have de novo (primary) or secondary AML (any WHO 2016 classification excluding acute promyelocytic leukemia) who have either comorbidities and/or advanced age (≥ 75 years) that preclude use of intensive induction chemotherapy as determined by the investigator.
4. Patients must be therapy-naïve (newly diagnosed)
5. Patients must have CD123-positive AML as confirmed by centralized flow cytometry (or immunohistochemistry [IHC]).
6. Patients with precedent MDS are eligible
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
8. Patients with previously untreated AML (by the World Health Organization (WHO) criteria, i.e. >/= 20% blasts). Prior biologic therapies (such as growth factors) and targeted therapies administered for the treatment of prior myelodysplastic syndrome are allowed (such as lenalidomide or luspatercept), with the exception of hypomethylating agents 5-azacytidine or decitabine. Patients must have been off such therapy for 1 week prior to entering this study and recovered from the toxic effects of that therapy, unless there is evidence of rapidly progressive disease. Hydroxyurea is permitted for control of counts prior to treatment.
9. Life expectancy of > 2 months in the Investigator's opinion
10. Creatinine ≤ 2.5 × upper limit of normal (ULN)
11. Adequate liver test parameters: total bilirubin < 2.5 × ULN (if disease related or secondary to Gilbert's disease, then total bilirubin < 3.5 mg/dL), aspartate aminotransferase (AST), and alanine aminotransferase (ALT) < 5 × ULN
12. Prothrombin time (PT) / international normalized ratio (INR) and partial thromboplastin time (PTT) < 2 × ULN
13. Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) may participate, provided they meet the following conditions:

    1. Must agree to use physician-approved contraceptive methods (e.g., abstinence, intrauterine device, oral contraceptive, double barrier device) throughout the study and for 3 months following the last dose of APVO436; and
    2. Must have a negative serum or urine pregnancy test within 7 days prior to beginning treatment on this study.
14. Males with female partners of child-bearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 3 months following the last dose of APVO436

Exclusion Criteria:

Subjects with any of the following will not be eligible for study participation:

1. Acute promyelocytic leukemia (APL) with t(15;17) translocation
2. Absolute peripheral blood myeloblast count greater than 20,000/mm3 - may receive hydroxyurea to reduce and control the myeloblast count down prior to and during the first week of the first cycle of treatment with study drug if necessary if deemed medically necessary and appropriate by the treating physician
3. Patients with active central nervous system (CNS) involvement by AML will be excluded. A lumbar puncture does not need to be performed unless there is clinical suspicion of CNS involvement per investigator judgement. Concurrent therapy for CNS prophylaxis or continuation of therapy for controlled CNS AML is allowed with the approval of the sponsor.
4. History of seizures
5. Prior solid organ transplant is acceptable provided the patient is on no immunosuppressive therapy.
6. Any therapy or experimental treatment for AML within 7 days of the first dose of study drug. The use of hydroxyurea is acceptable and does not exclude the patient.
7. Active, uncontrolled infection requiring systemic therapy. If the infection is controlled or has resolved, maintenance and/or prophylactic systemic antimicrobials are permitted.
8. Major surgery within 3 weeks prior to first dose of study drug
9. Known to be positive for HIV, hepatitis B virus surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C virus (HCV)
10. Uncontrolled hypertension, defined as blood pressure ≥ 140/90 mm Hg despite maximum medical intervention
11. History of congenital long QT syndrome or torsades de pointes
12. Pathologic bradycardia or heart block (excluding first degree heart block)
13. Prolonged baseline QTc, defined as QTcF (Fredericia correction) interval >480 msec (other correction formulas may be used for patients with bundle branch block or ventricular pacemaker)
14. History of ventricular arrhythmia (excluding PVCs)
15. Major surgery within 28 days prior to informed consent
16. Unstable angina pectoris within 28 days
17. Myocardial infarction and/or new ST elevation or depression or new Q wave on ECG within 6 months
18. Any history of stroke
19. Symptomatic congestive heart failure Class III or greater (New York Heart Association Functional Classification)
20. On full dose anti-coagulation defined as warfarin intended to raise the INR to 2-3
21. Major hemorrhagic event within 28 days requiring transfusion of packed red blood cells
22. Prior history of hypertensive crisis or hypertensive encephalopathy
23. Clinical evidence suggestive of central nervous system (CNS) involvement with leukemia unless a lumbar puncture was performed to confirm the absence of leukemic blasts in the cerebrospinal fluid (CSF)
24. Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
25. Any open wound
26. Pregnant and nursing subjects are excluded because the effects of APVO436 on a fetus or nursing child are unknown
27. Hydroxyurea is allowed prior to starting the study, and may be used for two weeks after dosing in Cycle 1 (e.g., Days 1-14 dosed with hydroxyurea)
28. Substance use disorder, psychiatric, cognitive, or any other condition that, in the opinion of the Investigator, would pose a risk to the patient's safety, may compromise the patient's ability to understand and comply with the protocol or provide informed consent, or interfere with the study evaluation, study participation, or follow-up
29. Any difficulty complying with protocol requirements that may increase the risk associated with study participation or study drug administration, or may cause a safety concern for the patient
30. Any uncontrolled medical condition, including but not limited to:
31. Uncontrolled metabolic disorders such as hypercalcemia
32. Any other active systemic malignancies. Exceptions: noninvasive non-melanoma skin cancer, in situ carcinoma, cervical intraepithelial neoplasia, and breast or prostate cancer that is well controlled with anti-hormonal therapy
33. Any current autoimmune disorder requiring immunosuppressive therapy with more than a replacement dose of corticosteroids (i.e., > 10 mg/day of prednisone or equivalent)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Safety - Incidence of Grade 3-4 AEs and SAEs | during first 28 to 35 days of treatment
  The cumulative incidence of Grade 3-4 AEs, and SAEs, and the incidence of AES of interest (≥Grade 2 CRS, ≥Grade 2 Infusion related reaction, ≥2 cardiac toxicity and ≥2 neurotoxicity as complications of CRS) for safety

SECONDARY OUTCOMES:
Efficacy - Incidence of composite CR (CR + CRi + CRh) | Patient will have assessment at the end of each Cycle (each Cycle is 28 days) up to 6 months
  Incidence of CR/CRi/CRh (composite CR rate) as a measure of efficacy within the confines of a Phase 1B study
Efficacy - Incidence of HSCT | Patient will have assessment after 1 year
  Incidence of HSCT post protocol therapy
Exploratory - LFS rate | up to 6 months
  Leukemia-free survival (LFS)
Exploratory - 1-year LFS rate | 1 year
  1-year LFS rate
Exploratory - 2-year LFS rate | 2 year
  2-year LFS rate
Exploratory - MRD burden | Patient will have assessment at the end of Cycle 1, 2 an 4 (each Cycle is 28 days) up to 6 months
  Post-protocol therapy (after 1 cycle, 2 cycles, and 4 cycles) MRD burden by MPFC